CLINICAL TRIAL: NCT00222118
Title: Promoting and Supporting Breastfeeding in Adolescents
Brief Title: Kansas University Teen Mothers Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR007773-01A2 (NIH); R01NR007773-01A2 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Pregnant Adolescents
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): intervention group
  Interventions: Other: intervention
- 2 (Other): Attention control
  Interventions: Behavioral: labor/birth preparation classes
- 3 (Other): Usual care
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: labor/birth preparation classes — prenatally, peer counselor/advanced practice nurse team, hospital visit, peer counselor telephone support for 4 weeks
  Arms: 2
Other: intervention — prenatal classes and phone calls from peer counselor, peer counselor/lactatin consultant, hospital visit, telephone support to 4 weeks postpartum
  Arms: 1
Other: usual care — no intervention
  Arms: 3

SUMMARY:
Breastfeeding initiation and duration in adolescent mothers.

DETAILED DESCRIPTION:
Randomized clinical trial to test the effects of a comprehensive prenatal, in-hospital, and postpartum education and support intervention on breastfeeding initiation and duration among teenage mothers. Experimental, attention control, and usual care groups are used to test the hypotheses. Drawing on the Theory of Planned Behavior and begun during the second trimester of pregnancy, the experimental condition uses a lactation consultant-peer counselor team to influence pregnant adolescents' beliefs and intentions about breastfeeding their newborns. The attention control (placebo) condition mimics the experimental condition, using an advanced practice nurse and peer counselor intervention team, and focuses on healthy pregnancy behaviors and labor/birth preparation. Teens in the two intervention groups attend two prenatal classes specific to their focus between the fourth and ninth month of pregnancy and receive telephone calls from a peer counselor. Teens in a usual care group receive no interventions beyond their standard prenatal care and education. After giving birth and still in the hospital, teens in the intervention groups receive a peer counselor phone call and visit. Breastfeeding teens in the experimental group also receive a breastfeeding counselor visit. After hospital discharge, breastfeeding teens from both intervention groups continue to receive peer counselor telephone support and, in the experimental condition, breastfeeding counselor phone calls for four weeks. Breastfeeding teens from all three groups complete short telephone interviews until six months after birth or until they stop breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-18 years
2. Adolescents intending to keep their newborns
3. 14 to 27 weeks of gestation
4. Ability to speak and read English
5. Possession or access to a telephone for study contact

Exclusion Criteria:

1. Multiple gestation pregnancy
2. Premature birth
3. Infant with cleft lip/palate, congenital heart defects, Down Syndrome, neural tube defects, or other conditions warranting the newborn's admission to neonatal intensive care
4. Subjects treated for significant complications during labor and birth that prohibit or delay breastfeeding beyond 48 hours or that have other conditions for which breastfeeding is contraindicated (e.g. HIV)

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome is breastfeeding initiation at hospital discharge. | hospital discharge

SECONDARY OUTCOMES:
Breastfeeding duration (in days) at 6 months postpartum | 6 months postpartum
Knowledge, attitudes, subjective norms, perceived behavioral control, and intentions regarding infant feeding prenatally | at enrollment, 36 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wambach, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States